CLINICAL TRIAL: NCT02743364
Title: Statin Therapy to Reduce the Risk of Recurrent Pancreatitis
Brief Title: Simvastatin in Reducing Pancreatitis in Patients With Recurrent, Acute or Chronic Pancreatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2016-00437; NCI-2016-00437 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00035; NCI2014-04-01 (Other: Northwestern University); NWU2014-04-01 (Other: DCP); N01CN00035 (NIH); P30CA060553 (NIH)
Record Dates: First submitted 2016-04-15; First posted 2016-04-19 (Estimated); Results first posted 2022-01-04 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-05

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (simvastatin) (Experimental): Patients receive simvastatin PO QD for 6 months.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Simvastatin
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD for 6 months.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo Administration — Given PO
  Arms: Arm II (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Simvastatin — Given PO
  Other Names: MK 733; Synvinolin; Zocor
  Arms: Arm I (simvastatin)

SUMMARY:
This randomized phase II trial studies how well simvastatin works in reducing pancreatitis (the inflammation of the pancreas) in patients with pancreatitis that occurs more than once (recurrent), has worsened quickly (acute), or has persisted or progressed over a long period of time (chronic). Simvastatin may decrease the inflammation of the pancreas by modulating the immune response responsible for inflammation. It is not yet known if simvastatin may be an effective treatment for pancreatitis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effect of a simvastatin intervention versus placebo on the change in secretin-stimulated peak bicarbonate concentration in the pancreatic fluid at 6 months post-treatment in patients with a history of at least two episodes of acute pancreatitis in the past 12 months.

SECONDARY OBJECTIVES:

I. To evaluate the effect of a simvastatin intervention versus placebo at 6 months from baseline (study visit

1) on: Ia. Change in the endoscopic ultrasound score (EUS). Ib. Change in serum and pancreatic fluid levels of cytokines, chemokines, and adhesion molecules.

Ic. Change in pancreatitis-related readmissions. Id. Change in quality of life score as measured by the Quality of Life (QLQ)-Core (C)30 and QLQ-Pancreatic modification (PAN)28(Chronic Pancreatitis [CP]).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive simvastatin orally (PO) once daily (QD) for 6 months.

ARM II: Patients receive placebo PO QD for 6 months.

After completion of study treatment, patients are followed up at 30, 60, and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* At least two episodes of acute pancreatitis in the past 12 months; acute pancreatitis is defined any 2 of the following: (1) typical upper abdominal pain; (2) elevation in serum amylase or lipase >= 3 times upper limit of normal; (3) features of acute pancreatitis on cross-sectional imaging
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 2,500/microliter
* Absolute neutrophil count >= 1,500/microliter
* Platelets >= 100,000/microliter
* Hemoglobin > 10 g/dL
* Total bilirubin =< 3.0 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x institutional ULN; patients whose AST/ALT levels normalize by screen 2 after an abnormal test will be included in the trial
* Creatinine < 1.5 mg/dL
* Women of child-bearing potential must have a confirmed negative pregnancy test result prior to enrollment
* The effects of simvastatin on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because statins are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately; it is not known whether simvastatin is excreted into human milk; however, a small amount of another drug in this class does pass into breast milk; because statins have the potential for serious adverse reactions in nursing infants, women who receive treatment with simvastatin should not breastfeed their infants
* Ability to understand and the willingness to sign a written informed consent document and medical release
* Willing and able to comply with trial protocol and follow-up

Exclusion Criteria:

* Prior or current use of statin medication, or current use of gemfibrozil, cyclosporine, danazol, lomitapide, verapamil, diltiazem, dronedarone, amiodarone, amlodipine, ranolazine, or strong cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors (e.g., itraconazole, ketoconazole, posaconazole, voriconazole, human immunodeficiency virus [HIV] protease inhibitors, boceprevir, telaprevir, erythromycin, clarithromycin, telithromycin, nefazodone, or cobicistat-containing products)
* History of chronic myopathy
* Current use of any other investigational agents
* History of adverse effects, intolerance, or allergic reactions attributed to compounds of similar chemical or biologic composition to simvastatin (i.e., other statin medications)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Women who are pregnant or breastfeeding; pregnant women are excluded from this study because simvastatin is a lipid-lowering agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with simvastatin, breastfeeding should be discontinued if the mother is treated with simvastatin
* Presence of gallstones and hypertriglyceridemia (level greater than 800 mg/dl) that requires medical or surgical intervention; note: we will include patients who had an independent episode of pancreatitis after a cholecystectomy, but exclude patients who are candidates for cholecystectomy
* History of pancreatic adenocarcinoma (at any time)
* History of active malignancy in the past 2 years (excluding basal/squamous cell skin cancer or prostate cancer with a Gleason score 6 or less)
* Known active infection with HIV
* Concurrent illness, such as known psychiatric disorders or substance abuse (i.e., average alcohol consumption of more than 5 drinks per day), which in the opinion of the investigators would compromise either the patient or the integrity of the data
* Laboratory (lab) results do not meet inclusion criteria
* Recurrent pancreatitis episode is iatrogenic (endoscopic retrograde cholangiopancreatography [ERCP] induced)
* Advanced chronic pancreatitis as determined by the following criteria: EUS score greater than 6, calcifications in combination with atrophy and/or dilation of >= 5 mm, or evidence of advanced chronic pancreatitis by computed tomography (CT) or magnetic resonance imaging (MRI) results in the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc T Goodman, Principal Investigator — Northwestern University
Locations (5):
- United States (5):
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Southern California Permanente Medical Group, Pasadena, California
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Simvastatin) | Arm II (Placebo)
Started | 6 | 2
Completed | 6 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients who have had at least two episodes of pancreatitis within the past 12 months.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Simvastatin) | Arm II (Placebo) | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (12.9) | 35.0 (11.3) | 43.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Bicarbonate Concentration, Measured Using Endoscopic Pancreatic Function Test (ePFT)
Description: Change in peak bicarbonate level (mmol/l) from baseline up to 6 months. Decreased peak bicarbonate concentration indicates worsening pancreatic function.
Time Frame: Baseline to up to 6 months
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Arm I (Simvastatin) | Arm II (Placebo)
Number analyzed (Participants) | 6 | 2
mmol/l | -8.20 (22.7) | 5.50 (0.707)

2. Secondary Outcome: Change in the Endoscopic Ultrasound Score (EUS)
Description: Change in EUS score (0-96) from baseline to up to 6 months. EUS Score is a measure of pancreatitis by the presence or absence of nine ductal and parenchymal criteria for CP: hyperechoic foci, hyperechoic strands, cysts, lobularity, calcifications, hyperechoic duct margins, visual side branches, main pancreatic duct dilation, and main pancreatic duct irregularity, which sum to a score ranging from 0 to 96. Presence of 6 or more standard criteria indicates advanced chronic pancreatitis. A positive score indicates an improvement. A negative score indicates a reduction.
Time Frame: Baseline to up to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Simvastatin) | Arm II (Placebo)
Number analyzed (Participants) | 6 | 2
score on a scale | 0.500 (1.38) | 0.500 (0.707)

3. Secondary Outcome: Serum and Pancreatic Secretions
Description: Expression of three biomarkers, HGF (hepatocyte growth factor), Resistin, and FASL (Fas ligand) in fluorescent intensity (arbitrary units), as an estimate of immune analyte concentration.
Time Frame: Baseline and 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: median fluorescent intensity
Arm/Group | Arm I (Simvastatin) | Arm II (Placebo)
Number analyzed (Participants) | 6 | 2
median fluorescent intensity
  Baseline HGF | 5.72 [5.20 to 6.22] | 7.13 [6.25 to 8.01]
  6 month HGF | 5.76 [5.29 to 6.23] | 5.99 [5.18 to 6.80]
  Baseline Resistin | 13.79 [12.99 to 14.60] | 12.39 [11.93 to 12.86]
  6 month Resistin | 12.94 [11.83 to 14.05] | 12.45 [11.81 to 13.10]
  Baseline FASL | 4.99 [4.67 to 5.30] | 4.83 [4.65 to 5.02]
  6 month FASL | 4.83 [4.48 to 5.18] | 4.82 [4.62 to 5.02]

4. Secondary Outcome: Pancreatitis-related Readmissions
Description: Number of participants with pancreatitis-related hospital readmissions.
Time Frame: Baseline to up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Simvastatin) | Arm II (Placebo)
Number analyzed (Participants) | 6 | 2
Participants | 5 | 1

5. Secondary Outcome: Change in Health-related Quality of Life.
Description: Change in health-related quality of life scores (1-100) from baseline to up to 6 months measured by the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 and EORTC QLQ-PAN28(CP) scores. A positive value indicates improvement and a negative value indicates reduction.
Time Frame: Baseline to up to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Simvastatin) | Arm II (Placebo)
Number analyzed (Participants) | 6 | 2
score on a scale
  Physical Functioning | 5.6 (6.6) | 6.7 (9.4)
  Role Functioning | 30.6 (35.6) | 25.0 (35.4)
  Cognitive Functioning | 2.8 (6.8) | 16.7 (23.6)
  Social Functioning | 22.2 (36.0) | 8.3 (35.4)
  Fatigue | -22.2 (35.1) | -50.0 (39.3)
  Pain | -8.3 (36.1) | -25.0 (35.4)
  Insomnia | -22.2 (50.2) | -33.3 (47.1)
  Overall | 19.4 (19.5) | 33.3 (0)

ADVERSE EVENTS:
Time Frame: AEs collected from the time informed consent was signed and baseline procedures were completed through 90 days post-intervention. In total AEs collected for a period of 9 months.
Arm/Group | Arm I (Simvastatin) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 5/6 | 1/2
Other Adverse Events (participants affected / at risk) | 5/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Simvastatin) (N=6) | Arm II (Placebo) (N=2)
Pancreatitis (Gastrointestinal disorders) | 5 (12) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Simvastatin) (N=6) | Arm II (Placebo) (N=2)
Abdominal Pain (Gastrointestinal disorders) | 5 (15) | 2 (3)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) — Appetite loss
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT02743364/Prot_SAP_000.pdf